CLINICAL TRIAL: NCT04249180
Title: Assessment of the Lived Experience of the Disease of the Patients Followed at the CHU of Gui de Chauliac for a Keratoconus and Their Habit of Eye Rubbing
Brief Title: Eye Rubbing and Keratoconus in Montpellier CHU
Acronym: Rub'Cornea
Status: Withdrawn | Type: Observational
Why Stopped: CPP
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0036
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Keratoconus
Keywords: primitive corneal ectasia; Ophthalmology; Eyes rubbing; Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluate the illness experience of patients with keratoconus as well as the rubbing habits of this population compared to the general population. To do this, the investigators used a questionnaire made by a Bordeaux team with questions on the experience of the patients' illness, their management and their friction habits

ELIGIBILITY:
Inclusion criteria:

- Having a keratonus at least in one eyes

Exclusion criteria:

- Refus to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient is having a keratoconus in at least one eye. It is a deases with a primitive corneal ectasia.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Assess whether eye rubbing is a risk factor for keratoconus | 1 day
  Assess whether eye rubbing is a risk factor for keratoconus

SECONDARY OUTCOMES:
Evaluate the habits of the population with a keratoconus | 1 day
  Evaluate the habits of the population with a keratoconus by a questionnaire completed by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Planells, Internship of ophthalmology, Principal Investigator — University Hospitals of Montpellier
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC